CLINICAL TRIAL: NCT04847180
Title: Study of the Antipodal Capsular Fold and Its Potential Role in Antero-inferior Glenohumeral Instability - Instabio
Brief Title: Study of the Antipodal Capsular Fold and Its Potential Role in Antero-inferior Glenohumeral Instability
Acronym: INSTABIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Ramsay santé (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ID-RCB : 2019-A00859-48
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Shoulder Capsulitis
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instability shoulder group (Experimental): Patients operated for an antero-inferior shoulder instability
  Interventions: Procedure: Biopsy
- Non instability shoulder group (Other): Patients without shoulder instability, operated for another reason.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — The biopsy will be performed at the level of the capsular fold located just above the area devoid of cartilage in the postero-superior region of the humeral head, near the area where Hill Sachs notches occur.

SUMMARY:
In schoulders instabilty, the soft tissue has not been the subject of histological studies, as has the "bare area" or zone devoid of cartilage, the exact role of which in glenohumeral biomechanics is unknown. This research is based on the hypothesis that the antipodal lesions are constant, underestimated and that an architectural disorganization at the capsulo-ligament level could contribute to the instability of the shoulder. The aim of this study is therefore to better characterize these lesions which could be the subject of a complementary stabilization procedure even in the absence of a humeral notch

DETAILED DESCRIPTION:
Surgery for unstable shoulders sometimes involves repairing lesions that promote instability. These lesions are identified on imaging before surgery and then during the operation, but they are macroscopically inconsistent on genuine unstable shoulders. While the importance of posterior capsuloligamentous structures (soft tissue) in antero-inferior stability has been the subject of biomechanical studies, the soft tissue has not been the subject of histological studies, as has the "bare area" or zone devoid of cartilage, the exact role of which in glenohumeral biomechanics is unknown. However, this research is based on the hypothesis that the antipodal lesions are constant, underestimated and that an architectural disorganization at the capsulo-ligament level could contribute to the instability of the shoulder. The aim of this study is therefore to better characterize these lesions which could be the subject of a complementary stabilization procedure even in the absence of a humeral notch.

ELIGIBILITY:
Inclusion Criteria:

Instability Group

* Patient, male or female, over 18 years old and up to 40 years old
* Patient operated for antero-inferior shoulder instability
* Subject affiliated or beneficiary of a social security scheme
* Patient having signed the free and informed consent comparativ group
* Patient, male or female, over 18 years old and up to 40 years old
* Patient operated for a reason other than unstable shoulder
* Subject affiliated or beneficiary of a social security scheme
* Patient having signed the free and informed cons

Exclusion Criteria:

* History of surgery on the affected shoulder
* Capsuloligamentous disease (Ehler Danlos)
* History of instability (dislocation, subluxation) in witnesses
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision;
* Pregnant, breastfeeding or parturient woman;
* Patient hospitalized without consent.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Capsule Aspect | during biopsy
  Normal capsule versus pathological capsule (abnormal capsule with disorganized framework, fragmented fibers, coiled )

CONTACTS AND LOCATIONS:
Overall Officials: Régis GUINAND, Dr, Principal Investigator — Clinique de l'Union - Ramsay-santé
Locations (1):
- Clinique de l'Union, Saint-Jean, France

IPD SHARING:
Plan to Share IPD: Undecided